CLINICAL TRIAL: NCT04012372
Title: Short-term Safety of ROSA Oligomineral Water in Healthy Serbian Infants
Brief Title: ROSA Oligomineral Water for Oral Hydration in 6-Month-Old Healthy Infants
Acronym: ROSAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Novi Sad, Faculty of Sport and Physical Education (Other)
Collaborators: Dom Zdravlja Nis (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 01-CC2019
Record Dates: First submitted 2019-07-04; First posted 2019-07-09 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Hydration
Keywords: Infants; Water; Safety

STUDY DESIGN:
Intervention Model Description: All participants will be allocated in an open-label manner to two randomly assigned ad libitum hydration regimens: first group will receive ROSA water for daily hydration, and second (control) group will receive other water of personal choice (including tap water)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ROSA water (Experimental): Ad libitum hydration with ROSA oligomineral water
  Interventions: Other: ROSA Water
- Control water (Active Comparator): Ad libitum hydration with other waters
  Interventions: Other: Control water

INTERVENTIONS:
Other: ROSA Water — Ad libitum hydration with ROSA oligomineral water
  Arms: ROSA water
Other: Control water — Ad libitum hydration with other waters
  Arms: Control water

SUMMARY:
The present study evaluates the safety of ROSA oligomineral water in 6-to-12-month old healthy children.

DETAILED DESCRIPTION:
Our study is designed as an open-label case-control interventional study that evaluates the safety of 28-day hydration with ROSA water in healthy infants aged 6-12 months. The participants are apparently healthy children breastfed or formula fed; minimal sample size (n = 52) was calculated according to 0.8 power to detect a significant difference in the prevalence of diarrhea (G*Power 3.1). Final group of participants will consist of sixty-five healthy male and female infants (we presume that 20% of participants will drop-out throughout the study). The stopping rules for participants include a refuse to participate in this research at any time and significant change of health status. All participants will be allocated in an open-label manner to two randomly assigned ad libitum hydration regimens: first group will receive ROSA water for daily hydration, and second (control) group will receive other water of personal choice (including tap water). All testing including parental diary of infant general status (e.g. daily amount of water consumed, number of stools per day, nutritional habits) and clinician-reported outcomes (e.g. body weight, clinical evaluation of hydration will be conducted at pre-administration (baseline) and at follow-up (after 28 days of administration). The study is entirely voluntary and the participants are free to stop participating at any time.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to 12 months
* Healthy children
* Doubled weight at 6 months
* Tripled weight at 12 months
* Feed with breast milk of milk formula

Exclusion Criteria:

* Any acute or chronic disease
* Unwillingness to return for follow-up analysis

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2019-07-20 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-10-07 (Actual)

PRIMARY OUTCOMES:
Daily amount of water consumed | Baseline vs. 28-days
  Monitor change in daily amount of water consumed

SECONDARY OUTCOMES:
Number of stools per day | Baseline vs. 28-days
  Monitor change in number of stools per day
Body weight | Baseline vs. 28-days
  Monitor change in body weight
Hydration status | Baseline vs. 28-days
  Monitor clinican-reported change in hydration status

CONTACTS AND LOCATIONS:
Overall Officials: Milorad Jerkan, MD, PhD, Principal Investigator — Dom Zdravlja Nis
Locations (1):
- Dom zdravlja Nis, Niš, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suh H, Kavouras SA. Water intake and hydration state in children. Eur J Nutr. 2019 Mar;58(2):475-496. doi: 10.1007/s00394-018-1869-9. Epub 2018 Nov 30. PMID 30506317
- [Background] Manz F. Hydration in children. J Am Coll Nutr. 2007 Oct;26(5 Suppl):562S-569S. doi: 10.1080/07315724.2007.10719659. PMID 17921466